CLINICAL TRIAL: NCT04687592
Title: Radiological and Functional Outcomes of Internal Fixation Methods for Vertical Femoral Neck Fractures in Young Adult Patients
Brief Title: Vertical Femoral Neck Fractures in Young Adult Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Thomas Magdi Labieb, resident at orthopedic department, Assiut University
Other Study IDs: Femoral Neck Fractures
Record Dates: First submitted 2020-11-15; First posted 2020-12-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Femoral Neck Fractures
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: reduction and fixation — * Reduction: one trial of closed reduction under anaesthesia and image control. Open reduction will be done by anterolateral or lateral approach if closed reduction failed
  * Fixation: internal fixation of the fracture by appropriate implant according to the fracture state

SUMMARY:
Does the current techniques of internal fixation of vertical neck fracture in young adult patients give a satisfactory radiological and functional outcome at one year follow up?

DETAILED DESCRIPTION:
* Displaced femoral neck fractures in young adults are most likely to result from high energy trauma that causes a vertically-oriented shearing injury through the femoral neck.
* The most descriptive classification used for femoral neck fractures in young patients is the Pauwels classification. As the degree of the femoral neck fracture line relative to the horizontal plane increases, the types differ (30 degrees type I, between 30 degrees and 50 degrees type II, 50 degrees type III), and the instability of the fracture.
* Greater fracture verticality contributes to greater difficulty in obtaining adequate stability to resist vertical shear forces around the hip, thereby resulting in ascending greater risk of complications such as nonunion and osteonecrosis despite a number of potential fixation strategies.
* The primary goals of surgery include preservation of the femoral head, avoidance of osteonecrosis, and achievement of a stable union.
* Fixation options include cannulated screws, sliding hip screw with or without an additional derotation screw,. among orthopedic trauma surgeons there is no consensus that a single fixation Option is superior for treating these injuries.

ELIGIBILITY:
Inclusion Criteria:

* Age of the patients from 20 to 50 years

  * Pauwel type III fractures
  * Recent fracture within one week

Exclusion Criteria:

* • Open fractures

  * Pathological or osteoporotic fractures.
  * Patient with comorbidities: D.M, renal patient, neurological deficits.
  * Patient associated with femoral head fractures or head impaction.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: adults patients with recent vertical femoral neck fracture
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
radiological and functional evaluation of the time and rate of union according harris hip score | one year
  The domains covered in Harris hip score are pain, function, absence of deformity, and range of motion. The pain domain measures pain severity and its effect on activities and need for pain medication.
  The function domain consists of daily activities (stair use, using public transportation, sitting, and managing shoes and socks) and gait (limp, support needed, and walking distance). Deformity takes into account hip flexion, adduction, internal rotation, and extremity length discrepancy. Range of motion measures hip flexion, abduction, external and internal rotation, and adduction .

REFERENCES:
- [Background] Macaulay W, Yoon RS, Parsley B, Nellans KW, Teeny SM; DFACTO Consortium. Displaced femoral neck fractures: is there a standard of care? Orthopedics. 2007 Sep;30(9):748-9. doi: 10.3928/01477447-20070901-08. PMID 17899921
- [Background] Bartonicek J. Pauwels' classification of femoral neck fractures: correct interpretation of the original. J Orthop Trauma. 2001 Jun-Jul;15(5):358-60. doi: 10.1097/00005131-200106000-00009. PMID 11433141
- [Background] Ye Y, Hao J, Mauffrey C, Hammerberg EM, Stahel PF, Hak DJ. Optimizing Stability in Femoral Neck Fracture Fixation. Orthopedics. 2015 Oct;38(10):625-30. doi: 10.3928/01477447-20151002-05. PMID 26488776
- [Background] Collinge CA, Mir H, Reddix R. Fracture morphology of high shear angle "vertical" femoral neck fractures in young adult patients. J Orthop Trauma. 2014 May;28(5):270-5. doi: 10.1097/BOT.0000000000000014. PMID 24096307
- [Background] Luttrell K, Beltran M, Collinge CA. Preoperative decision making in the treatment of high-angle "vertical" femoral neck fractures in young adult patients. An expert opinion survey of the Orthopaedic Trauma Association's (OTA) membership. J Orthop Trauma. 2014 Sep;28(9):e221-5. doi: 10.1097/BOT.0000000000000080. PMID 25148589